CLINICAL TRIAL: NCT03762421
Title: Evaluating a Multi-component Group Intervention for Improving Psychological Well-being of Trainee Civil Servants in Pakistan: a Randomised Controlled Study
Brief Title: Improving Psychological Well-being of Trainee Civil Servants in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Human Development Research Foundation, Pakistan (Other)
Collaborators: University of Liverpool (Other); Liverpool School of Tropical Medicine (Other); Civil Services Academy (CSA), Lahore (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-CS PM+
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Psychological Distress; Coping Skills; Well-being; Psychological Capital; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Fidelity of masking will be ensured by having assessors guess the condition of each participant at the end of each assessment to assess the contamination across intervention and control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosocial skills development workshops based on PM plus (Experimental): A number of psycho-social skills development workshops will be conducted for newly inducted civil servants, based on the problem management plus intervention. Problem Management Plus is a brief low-intensity, trans-diagnostic psychological intervention that helps with existing psychological problems as well as building resilience against future adversity. It addresses a range of psychological and practical problems that participants identify as relevant to their lives, including common mental health problems (WHO, 2016; Dawson, et al., 2015). The workshops will be integrated into the routine induction sessions for trainee civil servants.
  Interventions: Behavioral: Psycho-social skills development workshops based on PM plus
- Control Arm (Active Comparator): The control group will receive 5 routine training induction sessions.
  Interventions: Behavioral: Routine training induction sessions

INTERVENTIONS:
Behavioral: Psycho-social skills development workshops based on PM plus — 5 weekly, psycho-social skills development workshops will be conducted for newly inducted civil servants in groups, based on the problem management plus intervention. These workshops will be integrated into routine induction sessions of trainee civil servants. Workshop 1 orients participants to the intervention with motivational interviewing techniques to improve engagement, teaches the difference between technical and adaptive challenges, and trains participants in a basic stress management strategy. Workshop 2 addresses a participant-selected problem using problem-solving techniques and introduces behavioral activation. Workshops 3 and 4 support participants' continued application of problem solving, behavioral activation, and stress management and introduce strategies to strengthen social support networks whenever required. In Workshop 5, education about retaining intervention gains are provided and all learned strategies are reviewed.
  Arms: Psychosocial skills development workshops based on PM plus
Behavioral: Routine training induction sessions — The control group will receive 5 routine training induction sessions. These orientation sessions include lectures introduction to governance, public sector management, basic information technology, economics and public finance and official rules of procedure of the government of Pakistan. These lectures are held in a friendly and supportive environment.
  Arms: Control Arm

SUMMARY:
Political and civil instability in Pakistan has placed many segments of society under stress. A 5-session group intervention incorporating principles of stress management, problem solving, behavioural activation, peer-support and adaptive leadership has been developed and successfully piloted for business professionals working under stressful conditions in Pakistan. The aim of this study is to evaluate the effectiveness of an adapted version of the intervention in improving psychological well-being amongst a group of trainee civil servants in the country.

A two-arm single blind, randomised controlled trial of the group intervention will be conducted among trainee civil servants in Pakistan. The participants are newly inducted civil servants (n=240) undergoing a 6 months' induction training. The participants will be randomised on a 1:1 allocation ratio (120 in each arm), with the intervention arm receiving the group intervention integrated into their orientation sessions and the control arm receiving orientation sessions alone. Outcome assessments will be conducted immediately post-intervention and 3 months after the completion of the intervention. The primary outcomes will be change in the prevalence of psychological distress as measured by Patient Health Questionnaire-9 (PHQ-9) and improvement in coping strategies as measured by Brief Cope Questionnaire. Secondary outcomes include symptoms of anxiety (measured by Generalized Anxiety Disorder scale (GAD-7)), well-being (measured by WHO5 well-being index) and psychological capital (measured by Psychological Capital Questionnaire).

The primary analyses will be intent-to-treat consisting of all participants included, according to the groups in which they will be randomized. The primary analysis will involve comparing pre to post changes in prevalence of psychological distress and coping strategies of the participants randomly assigned to the two conditions, using Fisher's exact test. Primary analyses will be non-parametric tests; however sensitivity analyses will use parametric models such as linear and logistic regression to control for baseline values of the participants' characteristics.

Ethical principles of voluntary informed consent, maintaining anonymity and confidentiality, data management and storage will be followed.

ELIGIBILITY:
Inclusion Criteria:

* All newly inducted civil servants attending the CTP at the CSA, Lahore, which is a six months residential training course, and
* who give informed voluntary consent to take part in the study.

Exclusion Criteria:

* Participants having a physical health condition that does not allow them to attend the sessions will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The Patient Health Questionnaire-9 (PHQ-9) | One of the primary end points is the prevalence of psychological distress at 3 months post intervention
  One of the primary outcomes is change in the prevalence of psychological distress as measured by PHQ-9 in the intervention arm as compared to the control arm. The 9-item Patient Health Questionnaire (PHQ-9), incorporates DSM-IV depression diagnostic criteria with other key major depressive symptoms (Kroenke et al, 2001). Participants rate their responses on a 4-point Likert scale ranging from not at all to nearly every day. The PHQ-9 total severity score ranges from 0 to 27. Higher score represents high psychological distress. The PHQ-9 has been validated in the Urdu language, showing adequate sensitivity and specificity (Husain et al 2006) and has been used in recent studies in KP (Rahman et al, 2016).
Brief COPE | Another primary end point is the improvement in coping strategies at 3 months post intervention
  Another primary outcome is improvement in coping strategies measured by Brief COPE in the intervention arm as compared to the control arm. Brief COPE (Carver, 1997) is used to assess state coping (the way people cope with a specific stressful situation) and trait coping (the usual way people cope with stress in everyday life). It consists of 14 subscales i.e. active coping, planning, positive reframing, acceptance, humour, religion, use of emotional support, use of instrumental support, self-distraction, denial, venting, substance use, behavioral disengagement, and self-blame, with two items per sub-scale. The standard is to use sub-scale score. The score on each subscales ranges from 2 to 8. Higher score represents that person using the specific coping style a lot. Cronbach's alphas for the Brief COPE sub-scales range from 0.50 to 0.90 (Mayer, 2001).

SECONDARY OUTCOMES:
Psychological Capital Questionnaire (PCQ) | The secondary outcome data will be collected at 1 week post intervention and at 3 months post intervention
  Psychological capital will be measured using the Psychological Capital Questionnaire (PCQ) 12 items version (Avey et al, 2007). The PCQ-12 measures psychological capital across four domains (hope-4 items, optimism-2 items, resilience -3 items and self-efficacy-3 items). The participants rate their responses on 6 point likert scale. The total score ranges from 12-72. Higher scores represents higher psychological capital.
Generalized Anxiety Disorder -7 scale (GAD-7) | The secondary outcome data will be collected at 1 week post intervention and at 3 months post intervention
  GAD-7 will be used to measure anxiety (Spitzer et al, 2006) in the study sample. GAD-7 is based on the Diagnostic and Statistical Manual of Mental Disorders Version IV (DSM IV) diagnostic criteria for generalised anxiety disorder, and has 7 items. Each item is scored on a likert scale from 0 to 3, generating a maximum score of 21. High score represents presence of anxiety symptoms.
WHO-5 well-being index (WHO-5) | The secondary outcome data will be collected at 1 week post intervention and at 3 months post intervention
  Well-being will be measured by WHO 5 Well-being index (Topp, et al, 2015). WHO-5 is a short and generic global rating scale measuring subjective well-being, the respondent is asked to rate how well each of the 5 statements applies to him or her when considering the last 14 days. The instrument will be administered to study participants at 3 months post intervention to rate their subjective well being in last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). The raw score ranges from 0 (absence of well-being) to 25 (maximal well-being). Scores are then converted to a percentage scale from 0 (absent) to 100 (maximal). Higher scores represent greater psychological well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Development Research Foundation, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad S, Hussain S, Shah FS, Akhtar F. Urdu translation and validation of GAD-7: A screening and rating tool for anxiety symptoms in primary health care. J Pak Med Assoc. 2017 Oct;67(10):1536-1540. PMID 28955070
- [Background] Ahmer S, Faruqui RA, Aijaz A. Psychiatric rating scales in Urdu: a systematic review. BMC Psychiatry. 2007 Oct 26;7:59. doi: 10.1186/1471-244X-7-59. PMID 17963494
- [Background] Bolton P, Bass J, Neugebauer R, Verdeli H, Clougherty KF, Wickramaratne P, Speelman L, Ndogoni L, Weissman M. Group interpersonal psychotherapy for depression in rural Uganda: a randomized controlled trial. JAMA. 2003 Jun 18;289(23):3117-24. doi: 10.1001/jama.289.23.3117. PMID 12813117
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Chisholm D, Sweeny K, Sheehan P, Rasmussen B, Smit F, Cuijpers P, Saxena S. Scaling-up treatment of depression and anxiety: a global return on investment analysis. Lancet Psychiatry. 2016 May;3(5):415-24. doi: 10.1016/S2215-0366(16)30024-4. Epub 2016 Apr 12. PMID 27083119
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Goetzel RZ, Ozminkowski RJ, Sederer LI, Mark TL. The business case for quality mental health services: why employers should care about the mental health and well-being of their employees. J Occup Environ Med. 2002 Apr;44(4):320-30. doi: 10.1097/00043764-200204000-00012. PMID 11977418
- [Background] Husain N, Gater R, Tomenson B, Creed F. Comparison of the Personal Health Questionnaire and the Self Reporting Questionnaire in rural Pakistan. J Pak Med Assoc. 2006 Aug;56(8):366-70. PMID 16967789
- [Background] Jenkins R. Sex differences in minor psychiatric morbidity. Psychol Med Monogr Suppl. 1985;7:1-53. doi: 10.1017/s0264180100001788. PMID 3875115
- [Background] Jenkins R, Harvey S, Butler T, Thomas RL. Minor psychiatric morbidity, its prevalence and outcome in a cohort of civil servants--a seven-year follow-up study. Occup Med (Lond). 1996 Jun;46(3):209-15. doi: 10.1093/occmed/46.3.209. PMID 8695773
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Mirza I, Jenkins R. Risk factors, prevalence, and treatment of anxiety and depressive disorders in Pakistan: systematic review. BMJ. 2004 Apr 3;328(7443):794. doi: 10.1136/bmj.328.7443.794. PMID 15070634
- [Background] Patel V, Weiss HA, Chowdhary N, Naik S, Pednekar S, Chatterjee S, De Silva MJ, Bhat B, Araya R, King M, Simon G, Verdeli H, Kirkwood BR. Effectiveness of an intervention led by lay health counsellors for depressive and anxiety disorders in primary care in Goa, India (MANAS): a cluster randomised controlled trial. Lancet. 2010 Dec 18;376(9758):2086-95. doi: 10.1016/S0140-6736(10)61508-5. Epub 2010 Dec 13. PMID 21159375
- [Background] Rahman A, Hamdani SU, Awan NR, Bryant RA, Dawson KS, Khan MF, Azeemi MM, Akhtar P, Nazir H, Chiumento A, Sijbrandij M, Wang D, Farooq S, van Ommeren M. Effect of a Multicomponent Behavioral Intervention in Adults Impaired by Psychological Distress in a Conflict-Affected Area of Pakistan: A Randomized Clinical Trial. JAMA. 2016 Dec 27;316(24):2609-2617. doi: 10.1001/jama.2016.17165. PMID 27837602
- [Background] Rahman A, Malik A, Sikander S, Roberts C, Creed F. Cognitive behaviour therapy-based intervention by community health workers for mothers with depression and their infants in rural Pakistan: a cluster-randomised controlled trial. Lancet. 2008 Sep 13;372(9642):902-9. doi: 10.1016/S0140-6736(08)61400-2. PMID 18790313
- [Background] Rahman A, Riaz N, Dawson KS, Usman Hamdani S, Chiumento A, Sijbrandij M, Minhas F, Bryant RA, Saeed K, van Ommeren M, Farooq S. Problem Management Plus (PM+): pilot trial of a WHO transdiagnostic psychological intervention in conflict-affected Pakistan. World Psychiatry. 2016 Jun;15(2):182-3. doi: 10.1002/wps.20312. No abstract available. PMID 27265713
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Steel Z, Marnane C, Iranpour C, Chey T, Jackson JW, Patel V, Silove D. The global prevalence of common mental disorders: a systematic review and meta-analysis 1980-2013. Int J Epidemiol. 2014 Apr;43(2):476-93. doi: 10.1093/ije/dyu038. Epub 2014 Mar 19. PMID 24648481
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Whiteford HA, Degenhardt L, Rehm J, Baxter AJ, Ferrari AJ, Erskine HE, Charlson FJ, Norman RE, Flaxman AD, Johns N, Burstein R, Murray CJ, Vos T. Global burden of disease attributable to mental and substance use disorders: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Nov 9;382(9904):1575-86. doi: 10.1016/S0140-6736(13)61611-6. Epub 2013 Aug 29. PMID 23993280
- [Background] Whiteford HA, Ferrari AJ, Degenhardt L, Feigin V, Vos T. The global burden of mental, neurological and substance use disorders: an analysis from the Global Burden of Disease Study 2010. PLoS One. 2015 Feb 6;10(2):e0116820. doi: 10.1371/journal.pone.0116820. eCollection 2015. PMID 25658103
- [Background] Luthans, F., Avolio, B. J., Avey, J. B., & Norman, S. M. (2007). Positive psychological capital: Measurement and relationship with performance and satisfaction. Personnel psychology, 60(3), 541-572.
- [Background] Harnois G, Gabriel P, World Health Organization., 2000. Mental health and work: impact, issues and good practices.
- [Background] Heifetz R, Grashow A, Linsky M.,2009. The Practice of Adaptive Leadership: Tools and Tactics for Change your Organization and the World. Boston, MA: Harvard Business Review Press.
- [Background] Luthans, F., & Youssef, C. M. (2004). Human, social, and now positive psychological capital management: Investing in people for competitive advantage.